CLINICAL TRIAL: NCT00277693
Title: Protective Mechanisms of Aldosterone Antagonists and Their Effects on Cardiovascular Damage in Chronic Renal Failure: Clinical and Experimental Studies
Brief Title: Cardiovascular Protective Effect of Spironolactone in Hemodialysis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de los Andes, Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1040338
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2006-01-16 (Estimated); Status verified 2005-12

CONDITIONS: Hemodialysis
Keywords: hemodialysis; aldosterone; heart failure; spironolactone
MeSH Terms: conditions — Heart Failure | interventions — Spironolactone; Pharmaceutical Preparations

INTERVENTIONS:
Drug: Spironolactone (drug)

SUMMARY:
The purpose of the present study is to determine if spironolactone is safe and effective in the treatment of cardiovascular complications in hemodialysis patients.

DETAILED DESCRIPTION:
Cardiovascular complications are common in dialysis patients and comprise up to 50% of deaths in end-stage renal disease population. Hypertension and left ventricle hypertrophy occur in more than 70% of patients undergoing long-term hemodialysis therapy, and both contributes to mortality and morbidity.Recent clinical trials in chronic heart failure and post miocardial infarct heart failure patients have demonstrated a beneficial effect of a mineralocorticoid receptor blocker spironolactone, in adittion to standard therapy (RALES AND EPHESUS studies). The aim of the present study is to evaluate spironolactone treatment in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

chronic hemodialysys (> 3 months) anuria (diuresis <200 mL/day) -

Exclusion Criteria:

Liver failure Insulin dependent diabetes Treatment with adrenergic beta blockers or agonists Treatment with converting-enzime blocker or angiotensin receptor antagonists Cancer

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Luis F Michea, MD PhD, Study Chair — Faculty of Medicine, University Los Andes
Locations (1):
- Clinica Davila, Santiago, Santiago Metropolitan, Chile

REFERENCES:
- [Background] Michea L, Vukusich A, Gonzalez M, Zehnder C, Marusic ET. Effect of spironolactone on K(+) homeostasis and ENaC expression in lymphocytes from chronic hemodialysis patients. Kidney Int. 2004 Oct;66(4):1647-53. doi: 10.1111/j.1523-1755.2004.00931.x. PMID 15458462
- [Derived] Hasegawa T, Nishiwaki H, Ota E, Levack WM, Noma H. Aldosterone antagonists for people with chronic kidney disease requiring dialysis. Cochrane Database Syst Rev. 2021 Feb 15;2(2):CD013109. doi: 10.1002/14651858.CD013109.pub2. PMID 33586138